CLINICAL TRIAL: NCT01634256
Title: A Human Trial to Evaluate the Efficacy and Safety of Fermented Turmeric in Subjects Showing Mild Hepatic Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INs-LF-CURCUMA
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Mild Hepatic Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fermented turmeric (Experimental)
  Interventions: Dietary Supplement: Fermented turmeric
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo(3.0g/day)
  Arms: Placebo
Dietary Supplement: Fermented turmeric — Fermented turmeric(3.0g/day)
  Arms: Fermented turmeric

SUMMARY:
The investigators performed a double-blind parallel study in a group of showing mild hepatic injury subjects who were given Fermented turmeric over a period of 12 weeks. The investigators measured liver function parameters , including ALT(Alanine Transaminase), AST(Aspartate Transaminase), ALP(Alkaline Phosphatase), γ-GT(Gamma-Glutamyl Transferase), and serum bilirubin, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-70 years old
* Mild hepatic injury as indicated by ALT(Alanine Transaminase) level ≥ 40
* Able to give informed consent

Exclusion Criteria:

* Allergy or hypersensitivity to any of the ingredients in the test products
* History of reaction to any of the experimental products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* Carriers of viral hepatitis (type B and C)
* History of underlying Esophageal varices, hepatic encephalopathy, ascites(past 12 months)
* Participation in other clinical trials within the past 2 months
* Patients with acute hepatitis (type B and C)
* History of underlying cirrhosis and liver cancer
* History of underlying biliary diseases such as jaundice or gallstones
* History of underlying kidney disease such as Chronic renal failure or nephrotic syndrome
* Pregnant, planning to become pregnant, or breast-feeding
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Wook Kim, MS, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Kim SW, Ha KC, Choi EK, Jung SY, Kim MG, Kwon DY, Yang HJ, Kim MJ, Kang HJ, Back HI, Kim SY, Park SH, Baek HY, Kim YJ, Lee JY, Chae SW. The effectiveness of fermented turmeric powder in subjects with elevated alanine transaminase levels: a randomised controlled study. BMC Complement Altern Med. 2013 Mar 8;13:58. doi: 10.1186/1472-6882-13-58. PMID 23497020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 19 to 70 years, ALT levels ≥ 40IU/L subjects.
Groups:
- Fermented Turmeric: Fermented turmeric(3times/day, 6capsules/day, 3g/day) for 12weeks
  Fermented curcuma : Powdered Curcuma longa L., was produced through the fermentation of Aspergillus oryzae to 25 ˚ C for 36 hours.
- Placebo: Placebo(3times/day, 6capsules/day, 3g/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with Fermented turmeric.
Period: Overall Study
Arm/Group | Fermented Turmeric | Placebo
Started | 30 | 30
Completed | 26 | 22
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fermented Curcuma | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.03 (8.53) | 36.17 (7.42) | 37.60 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Changes in ALT(Alanine Transaminase)
Description: ALT was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Fermented Turmeric: Oral intake Fermented turmeric (3.0g/day) for 12weeks.
- Placebo: Oral intake placebo(3.0g/day) for 12weeks
Arm/Group | Fermented Turmeric | Placebo
Number analyzed (Participants) | 26 | 22
IU/L
  Pre | 61.08 (25.10) | 55.68 (15.09)
  Post | 44.92 (15.47) | 53.82 (26.27)

2. Secondary Outcome: Changes in AST(Aspartate Transaminase)
Description: AST was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fermented Turmeric | Placebo
Number analyzed (Participants) | 26 | 22
IU/L
  Pre | 36.27 (13.80) | 35.59 (8.82)
  Post | 27.96 (7.96) | 34.77 (10.87)

3. Secondary Outcome: Changes in ALP(Alkaline Phosphatase)
Description: ALP was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fermented Turmeric | Placebo
Number analyzed (Participants) | 26 | 22
IU/L
  Pre | 85.04 (19.33) | 71.73 (13.47)
  Post | 80.04 (21.98) | 68.95 (13.21)

4. Secondary Outcome: Changes in γ-GT(Gamma-Glutamyl Transferase)
Description: γ-GT was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fermented Turmeric | Placebo
Number analyzed (Participants) | 26 | 22
IU/L
  Pre | 86.31 (71.49) | 104.2 (69.00)
  Post | 66.96 (45.63) | 100.77 (68.36)

5. Secondary Outcome: Changes in Serum Bilirubin
Description: serum bilirubin was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fermented Turmeric | Placebo
Number analyzed (Participants) | 26 | 22
mg/dL
  Pre | 0.98 (0.46) | 0.89 (0.28)
  Post | 0.88 (0.38) | 0.84 (0.26)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Groups:
- Fermented Curcuma: Oral intake fermented curcuma (3.0g/day) for 12weeks.
Arm/Group | Fermented Curcuma | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No